CLINICAL TRIAL: NCT03092557
Title: A Pilot Study of a New Ultrasonographic Tool to Assess Regional Pulmonary Strain in Patients Under General Anesthesia
Brief Title: A New Ultrasonographic Tool to Assess Regional Pulmonary Strain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Centre hospitalier de l'Université de Montréal (CHUM) (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 16.386
Record Dates: First submitted 2017-03-12; First posted 2017-03-28 (Actual); Last update posted 2017-10-30 (Actual); Status verified 2017-10

CONDITIONS: Ventilator-Induced Lung Injury; Mechanical Ventilation Complication
MeSH Terms: conditions — Ventilator-Induced Lung Injury

STUDY DESIGN:
Intervention Model Description: Prospective, interventional, cohort study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Determination of local pleural strain (Experimental): Patients will receive four different tidal volumes in random order (6 mL/kg, 8 mL/kg, 10 mL/kg, 12 mL/kg).
  Interventions: Other: Determination of local pleural strain

INTERVENTIONS:
Other: Determination of local pleural strain — For each tidal volume, the local pleural strain will be determined over three consecutive respiratory cycles at four predetermined sites using lung ultrasonography.

SUMMARY:
This study is designed to assess the feasibility of the measurement of local pleural strain at 4 different anatomical sites.

The secondary objectives of the study are:

* To assess intra- and inter-observer variability in the measurement of local pleural strain
* To identify the strain parameters demonstrating the most clinically relevant and the most significant correlation with a change in tidal volume

Hypothesis: The analysis of lung ultrasonographic sequences using speckle-tracking allows the determination of local pleural strain in 4 predetermined pulmonary areas.

DETAILED DESCRIPTION:
Mechanical ventilation is frequently used in the operating room and the intensive care settings. Although essential in many cases, mechanical ventilation can be responsible for ventilator-induced lung injury (VILI). The relationship between mechanical ventilation and VILI has been clearly demonstrated in animals and is highly suspected in humans. The putative mechanism responsible for VILI is excessive pulmonary strain or overdistension. Frequently observed in mechanically ventilated patients, the presence of a severe pre-existing pulmonary disease can increase the risk of overdistension. The development of a tool allowing early detection of pulmonary overdistension would represent a great asset in the prevention of VILI by allowing safer adjustments of mechanical ventilation parameters. Ultrasonographic imaging is a non-radiant, non-invasive technique already available in the intensive care setting. Already used for cardiac strain measurements, ultrasonography is a promising avenue to assess pulmonary strain.

This pilot study will aim to assess the feasibility of the measurement of local pleural strain in 4 predetermined pulmonary areas using ultrasonographic imaging.

Following the induction of general anesthesia and the patient's intubation, 4 different tidal volumes of 6 ml/kg, 8ml/kg, 10 ml/kg and 12 ml/kg will be studied. For each volume, images of the pleura will be made at 4 predetermined areas. The sites to be studied will be: the 4th intercostal space at the mid-clavicular line (left and right side), the 7th intercostal space at the posterior axillary line (left and right side). For each tidal volume, 3 consecutive respiratory cycles at each site will be recorded for subsequent analysis.

To assess intra- and inter-observer variability, for the 10 ml/kg tidal volume only, the examination will be immediately repeated by a second observer at the 4 predetermined sites. The first observer will also return to repeat the examination at the same sites.

Mechanical ventilation parameters will be standardized throughout the study as follows: volume-controlled ventilation, respiratory rate at 12 breaths per minute adjusted to obtain expired carbon dioxide (CO2) between 30 and 40 mm Hg, initial inspired oxygen fraction of 40% adjusted between 40% and 80% to obtain oxygen saturation ≥ 92% and positive end-expiratory pressure at 6 cm H2O. In the event of a desaturation (saturation inferior to 90%) despite an increase in inspired oxygen fraction, the study will be stopped and adjustments of mechanical ventilation parameters will be left to the attending anesthesiologist's discretion.

Lung ultrasonography will be performed by the principal investigator and a co-investigator using a Terason (Teratech Corporation, Burlington, MA) device and a 12L5 linear ultrasound probe. For each image, the probe will be oriented perpendicularly to the ribs and pleura with the pointer towards the participant's head. Depth will be adjusted in order to have the pleural line in the center of the screen. The beam's focal zone will be positioned at the level of the pleural line. A 12 megahertz (MHz) frequency will be used.

Using a reference ultrasonographic image, an experienced lung ultrasonographer will segment the pleura. From this image, an algorithm will define a region of interest which will be followed throughout the rest of the images of the video sequence. Thereafter, the algorithm will calculate the various components of pulmonary strain in relation to tidal volume. An experienced technician will visually validate the speckle-tracking.

ELIGIBILITY:
Inclusion Criteria:

* Patients with presumed healthy lungs undergoing elective surgery under general anesthesia requiring neuromuscular blocking agents and orotracheal intubation

Exclusion Criteria:

* Previous thoracic procedure (chest tube, thoracotomy, thoracoscopy)
* Pre-existing pulmonary disease (asthma, chronic obstructive pulmonary disease, lung fibrosis)
* Active or previous history of smoking
* Need for supplemental oxygen
* Abnormal pulmonary function tests (when available)
* Obesity (Body Mass Index superior to 30 kg/m2)
* Functional capacity inferior to 4 metabolic equivalent of task (METs)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2017-07-24 (Actual); Primary Completion 2017-10-26 (Actual); Study Completion 2017-10-26 (Actual)

PRIMARY OUTCOMES:
Feasibility of the measurement of local pleural strain using ultrasonography | At the end of study on Day 1
  Proportion of successfully analyzed lung ultrasonographic clips

SECONDARY OUTCOMES:
Intra-observer variability | At the end of study on Day 1
  Agreement and bias will be calculated according to Bland and Altman
Inter-observer variability | At the end of study on Day 1
  Agreement and bias will be calculated according to Bland and Altman
Maximal axial deformation | At the end of study on Day 1
  Increase from baseline in percentage
Maximal lateral deformation | At the end of study on Day 1
  Increase from baseline in percentage
Mean magnitude of shear deformation | At the end of study on Day 1
  Increase from baseline in percentage
Cumulative axial translation | At the end of study on Day 1
  Difference from baseline in millimeters
Cumulative lateral translation | At the end of study on Day 1
  Difference from baseline in millimeters

CONTACTS AND LOCATIONS:
Overall Officials: Martin Girard, MD, FRCPC, Principal Investigator — Centre hospitalier de l'Université de Montréal (CHUM)
Locations (1):
- Centre Hospitalier de l'Université de Montréal (CHUM), Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Girard M, Roy Cardinal MH, Chasse M, Garneau S, Cavayas YA, Cloutier G, Denault AY. Regional pleural strain measurements during mechanical ventilation using ultrasound elastography: A randomized, crossover, proof of concept physiologic study. Front Med (Lausanne). 2022 Sep 15;9:935482. doi: 10.3389/fmed.2022.935482. eCollection 2022. PMID 36186794